CLINICAL TRIAL: NCT04044040
Title: Symptom Screening With Targeted Early Palliative Care (STEP) for Patients With Advanced Cancer: A Pilot Trial
Brief Title: Symptom Screening With Targeted Early Palliative Care (STEP) for Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB ID 16-5590
Record Dates: First submitted 2019-07-24; First posted 2019-08-02 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: Palliative care; Symptom control; Quality of life; Satisfaction with care; Targeted referral
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptom screening with Targeted Early Palliative care (STEP) (Experimental): The experimental arm receives routine symptom screening at every outpatient visit; if symptoms are above a certain threshold, then a triggered email is sent to a triage nurse, who calls the patient to offer early referral to and follow-up by a symptom control and palliative care team.
  Interventions: Behavioral: Symptom screening with Targeted Early Palliative care (STEP)

INTERVENTIONS:
Behavioral: Symptom screening with Targeted Early Palliative care (STEP) — The experimental arm receives routine symptom screening at every outpatient visit; if symptoms are above a certain threshold, then a triggered email is sent to a triage nurse, who calls the patient to offer early referral to and follow-up by a symptom control and palliative care team.

SUMMARY:
Palliative care is defined as multidisciplinary care that increases quality of life (QOL) for patients with a life-threatening illness. Although it is known that patients with the most severe physical and psychological symptoms have the greatest need for palliative care, these patients are often not referred to palliative care services in a timely manner.

We have developed a system called STEP (Symptom screening with Targeted Early Palliative care) that identifies patients with high symptom burden in order to offer them timely access to palliative care. The investigators are conducting a single-arm trial at Princess Margaret Cancer Centre to determine the feasibility of a larger randomized trial of STEP versus usual care and to establish specific parameters for its planning.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) have shown when patients with advanced cancer were referred early to specialized palliative care teams, they had improved QOL, symptom control, and greater satisfaction with their cancer care. Such routine specialized palliative care intervention, while effective, may be challenging to enact broadly with widespread shortages of palliative care physicians. STEP systematically identifies patients with the greatest need, using symptom screening at every outpatient visit, with triage and targeted referral to palliative care. This could reduce resource use while directing care to the most vulnerable.

Patients will be recruited from Breast, Lung, Gastrointestinal, Genitourinary, and Gynecology medical oncology clinics. Consenting participants will complete questionnaires measuring outcomes of QOL, symptom control, depression, and satisfaction with care at recruitment, 2, 4 and 6 months. The objectives of the study are to assess the feasibility of conducting a larger phase III trial and to collect information to assist in trial planning and sample size calculation for such a trial. Feasibility criteria are: i) ≥100 patients accrued in 12 months; ii) ≥70% complete screening for ≥70% of visits; iii) ≥60% of those for whom a call is triggered meet at least once with the EPC team; iv) ≥60% complete measures at each endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of stage IV cancer (advanced); hormone-refractory for breast or prostate cancer; stage III or IV for lung cancer and pancreatic cancer; patients with stage III cancer and poor clinical prognosis, e.g. ovarian or esophageal cancer, will be included at the discretion of the oncologist
* ECOG performance status ≤ 2 (estimated by primary oncologist)
* Prognosis of >6 months (estimated by primary oncologist)
* Patient completes symptom screening in outpatient clinic electronically

Exclusion Criteria:

* Insufficient English literacy to complete questionnaires
* Inability of pass the cognitive screening test (SOMC - Short Orientation Memory Concentration test score <20 or >10 errors)
* Receiving specialized palliative care within the last 6 months prior to screening, per chart and patient statement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Patient Heath Related Quality of Life (HRQL) as measured by the FACIT-Sp. | 6 months after enrollment
  The FACIT-Sp encompasses the FACT-G (Functional Assessment of Cancer Therapy-General) and FACIT spiritual well-being subscale to measure physical, social/family, emotional, functional and existential well-being.

SECONDARY OUTCOMES:
Patient Heath Related Quality of Life (HRQL) as measured by the FACIT-Sp. | 2 and 4 months after enrollment
  The FACIT-Sp encompasses the FACT-G (Functional Assessment of Cancer Therapy-General) and FACIT spiritual well-being subscale to measure physical, social/family, emotional, functional and existential well-being. Scores range from 0-156 with higher scores indicating better quality of life.
Patient Heath Related Quality of Life (HRQL) as measured by the QUAL-E. | 2, 4 and 6 months after enrollment
  The QUAL-E (Quality of Life at the End of Life) measures quality of life domains including life completion, symptoms impact, relationship with health care provider, and preparation for end of life. Scores range from 21-105 with higher scores indicating better quality of life.
Symptom control | 2, 4 and 6 months after enrollment
  Symptom control is measured by the 11-item ESAS-r-CS (Edmonton Symptom Assessment System-revised plus constipation and trouble sleeping). All 11 items are summed for the ESAS-r-CS Total Distress Score (TDS), where higher scores indicate worse symptom burden.
Depression | 2, 4 and 6 months after enrollment
  Depression is measured by the Patient Health Questionnaire (PHQ-9). Scores range from 0-27 with higher scores indicating worse depression.
Patient satisfaction with care | 2, 4 and 6 months after enrollment
  Satisfaction with care is measured by the FAMCARE-P16 (Family Satisfaction with Cancer Scale modified for patients). Scores range from 16-80 with higher scores indicating higher satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Zimmermann, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmermann C, Pope A, Hannon B, Krzyzanowska MK, Rodin G, Li M, Howell D, Knox JJ, Leighl NB, Sridhar S, Oza AM, Prince R, Lheureux S, Hansen AR, Rydall A, Chow B, Herx L, Booth CM, Dudgeon D, Dhani N, Liu G, Bedard PL, Mathews J, Swami N, Le LW. Phase II Trial of Symptom Screening With Targeted Early Palliative Care for Patients With Advanced Cancer. J Natl Compr Canc Netw. 2021 Sep 7;20(4):361-370.e3. doi: 10.6004/jnccn.2020.7803. PMID 34492632